CLINICAL TRIAL: NCT05962424
Title: HNC: Human Neural Circuits Electrophysiology During Cognition
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Karl Deisseroth, Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 70198
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Disorder
MeSH Terms: conditions — Mental Disorders | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Ketamine (Experimental): Study participants will receive 0.5mg/kg of ketamine - one single infusion
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine is an FDA-approved dissociative anesthetic.
  Other Names: Ketalar

SUMMARY:
The purpose of this study is to understand how ketamine brings about dissociative symptoms.

DETAILED DESCRIPTION:
The goal of this proposed research is to record the effects of ketamine on brain activity to understand the changes that occur during antidepressant therapy and the side effect of dissociation. This research is designed to probe altered cognitive states associated with dissociation, depression, and other neuropsychiatric conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patient in clinical neuro inpatient units at Stanford Medical Center
* Age >18 years old
* Female participants are expected to use an effective method of birth control throughout the study which includes: hormonal methods (birth control pills, patches, injections, vaginal ring or implants), barrier methods (condom or diaphragm) used with spermicide, intrauterine device (IUD), or abstinence (no sex)

Exclusion Criteria:

* Lifetime psychotic disorder
* Pregnant or nursing females
* Prior adverse ketamine response
* Use of ketamine in past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dissociative events during ketamine infusion as assessed by CADSS (Clinician-Administered Dissociative State Scale) | up to 1 week
  The CADSS is an instrument for the measurement of dissociative symptoms. The CADSS comprises 23 subjective items and participant's responses are coded on a 5-point scale (0 = Not at all; 4 = Extreme). The higher the number on the CADSS, the more severe the symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Deisseroth, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No